CLINICAL TRIAL: NCT00416078
Title: Caregiver Psychoeducation and Support: Improving Outcomes in AD/ADRD
Brief Title: Online Caregiver Psychoeducation and Support for Alzheimer's
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 05-107
Record Dates: First submitted 2006-12-22; First posted 2006-12-27 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Alzheimer's Disease
Keywords: technology development and assessment; internet; randomized control trial
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- caregiver website support (Experimental): caregiver access to website support for 6 months embedded in one year of customary care
  Interventions: Behavioral: caregiver website support
- caregiver brief supportive phone calls (Active Comparator): caregiver brief supportive telephone calls for 6 months embedded in one year of customary care
  Interventions: Behavioral: caregiver brief supportive phone calls

INTERVENTIONS:
Behavioral: caregiver website support — caregiver access to website support for 6 months embedded in one year of customary care
  Arms: caregiver website support
Behavioral: caregiver brief supportive phone calls — caregiver brief supportive telephone calls for 6 months embedded in one year of customary care
  Arms: caregiver brief supportive phone calls

SUMMARY:
This study is piloting an internet-based intervention to provide support for caregivers of VA patients with Alzheimer's disease or related memory difficulties (ADRD). Veterans with a clinical diagnosis of ADRD and their caregiver/relatives will be randomized to receive one of two interventions: (1) customary care (cc) and access to an intensive, interactive online education and support website intervention for 6 months, or (2) cc and monthly brief telephone calls with project staff for six month. It is hypothesized that participation in the intensive intervention will result in a reductions in patient problematic behavior and caregiver responses to it, reduced caregiver burden and depression, and improved medication adherence at the end of treatment, and more patients remaining at home through the 12 months post-randomization period..

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive brain disease resulting in cognitive and functional decline. While some pharmacological agents and behavioral programs are now available to slow the rate of decline, there is no cure. Caregivers, who typically are the female spouses or daughters of afflicted individuals, must confront both the deterioration of a loved one, and that person's need for increasingly demanding care. Caregivers tend to experience high levels of depression, anxiety, and burden. Data suggest that providing education, social support, and ongoing professional consultation to families involved in the care of a relative with AD results in improvement in caregiver psychological status, and sometimes even slows the functional decline of the patient.

Recent technological advancements in video conferencing, online communication, and streaming audio/video presentations, which are increasingly easy to use and gaining widespread acceptance among mental health professionals as well as the public, have given rise to a great deal of interest in telemedicine and telepsychiatry. This study tested an Internet-based family intervention for AD that relatives can access from their homes with ease, and at no cost. In addition to improving patient outcomes through instruction of effective behavioral management, we proposed that participation in an Internet program would also reduce caregiver depression and burden. Fifty-three veterans with a clinical diagnosis of AD and their caregiver/relatives were randomized to receive one of two interventions: (1) customary care (cc) and access to an intensive, interactive online education and support website intervention for 6 months, or (2) cc and monthly brief telephone calls with project staff for 6 months. We hypothesized that, at the end of the active intervention, participation in the intensive intervention would result reduced patient problematic behavior, caregiver burden, depression, and negative responses to problematic patient behaviors, as well as improved patient medication compliance. At 12 month follow-up, we hypothesized access to the online program would result in more patients remaining at home. The overriding longterm project objective was to develop an effective online education and support program for caregivers of patients with AD that can be manualized, replicated, and disseminated to other clinical and research centers, within both the VA health care system and the community, to enhance the efficiency and effectiveness of psychosocial treatment in AD.

ELIGIBILITY:
Inclusion Criteria:

* Patient living in community and ambulatory
* Patient has diagnosis of Alzheimer's disease
* Patient age 50-95
* Caregiver age 18-90
* Patient currently under treatment for Alzheimer's disease
* Patient and caregiver reside within 2 hours of Los Angeles
* Caregiver has home internet access
* Patient has close contact with caregiver

Exclusion Criteria:

* Patient lives in residential setting
* No family contact
* Acute illness or chronic disease in patient or caregiver
* Patient or caregiver plans to leave area within the year

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-08; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore J. Hahn, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States

REFERENCES:
- [Result] Hayden LJ, Glynn SM, Hahn TJ, Randall F, Randolph E. The use of Internet technology for psychoeducation and support with dementia caregivers. Psychol Serv. 2012 May;9(2):215-8. doi: 10.1037/a0027056. PMID 22662739
- [Derived] Gonzalez-Fraile E, Ballesteros J, Rueda JR, Santos-Zorrozua B, Sola I, McCleery J. Remotely delivered information, training and support for informal caregivers of people with dementia. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD006440. doi: 10.1002/14651858.CD006440.pub3. PMID 33417236

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregiver Website: relative access to website support for 6 months embedded in one year of customary care
- Caregiver Phone Calls: relative supportive telephone calls for six months embedded in one year of customary care
Period: Overall Study
Arm/Group | Caregiver Website | Caregiver Phone Calls
Started | 29 | 24
Completed | 18 | 16
Not Completed | 11 | 8
Not completed — Death | 3 | 4
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Caregiver Phone Calls: relative supportive telephone calls for six months embedded in one year customary care
- Total: Total of all reporting groups
Arm/Group | Caregiver Website | Caregiver Phone Calls | Total
Number analyzed (Participants) | 29 | 24 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] — Patient data presented here
  years | 78.69 (9.09) | 81.4 (6.6) | 79.92 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 22 | 19 | 41
Race/Ethnicity, Customized [Number; unit: patient participants]
  Caucasian | 20 | 19 | 39
  African-American | 6 | 4 | 10
  Hispanic | 1 | 1 | 2
  Unknown | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 29 | 24 | 53

OUTCOME MEASURES:

1. Secondary Outcome: Change in Caregiver Report of Patient Medication Adherence From Baseline
Description: Adherence to prescribed medication regimen rated by caregiver on a 1 (0%) to 5 (100%) scale. Higher scores indicate better adherence. Values in statistical table below are least square estimates, and thus may be slightly out-of-range of actual respondent choices on scale.
Time Frame: baseline to end-of-treatment (6 months)
Population: measure was added to study while in process
Measure: Least Squares Mean (Standard Error); unit: units on a 1-5 scale
Arm/Group | Caregiver Website | Caregiver Phone Calls
Number analyzed (Participants) | 9 | 16
units on a 1-5 scale
  at baseline | 4.63 (.47) | 4.06 (.42)
  at 6 months | 5.08 (.75) | 3.94 (.44)
Statistical Analysis 1: Comparison: Caregiver Website vs Caregiver Phone Calls; intent to treat; Test type: Superiority or Other; p = .65, Mixed Models Analysis — F test of time X group effect F(1,3)=.26

2. Primary Outcome: Change in Caregiver Burden From Baseline
Description: Total score on the Zarit Short Burden Scale, a 12 item instrument that utilizes a likert scale 1-5 rating of frequency. The range is 12 (never) to 60 (nearly always) wherein higher scores are more indicative of caregiver burden.
Time Frame: baseline to end-of-treatment (6 months)
Population: Data available for analyses vary due to missing data (lost to follow-up and deaths at different points in the protocol; incomplete forms)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Caregiver Website | Caregiver Phone Calls
Number analyzed (Participants) | 20 | 19
units on a scale
  baseline | 32.04 (1.95) | 28.59 (2.01)
  end of treatment | 32.52 (2.13) | 27.55 (2.19)
Statistical Analysis 1: Comparison: Caregiver Website vs Caregiver Phone Calls; intent to treat analysis; Test type: Superiority or Other; p = .51, Mixed Models Analysis — t test of differential change over time in the two groups t(30)=.67

3. Primary Outcome: Change in Frequency of Patient Problematic Behavioral Patterns From Baseline
Description: Total Score on the Frequency of Problematic Behaviors on the Revised Memory and Behavior Problem Checklist. The Revised Memory and Behavior Checklist is a 24 item instrument that measures the frequency of a behavior on a 0-4 likert scale wherein higher numbers indicate greater frequency. The range is 0-96.
Time Frame: baseline to end of treatment (6 months)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Caregiver Website | Caregiver Phone Calls
Number analyzed (Participants) | 20 | 20
units on a scale
  baseline | 30.69 (2.89) | 33.04 (2.99)
  end-of-treatment (6 months) | 33.28 (3.11) | 34.75 (3.27)
Statistical Analysis 1: Comparison: Caregiver Website vs Caregiver Phone Calls; intent to treat analysis; Test type: Superiority or Other; p = .79, Mixed Models Analysis — t test of differential change over time in the two groups t(29)=.27

4. Primary Outcome: Change in Caregiver Negative Reactions to Problematic Behavioral Patterns From Baseline
Description: Total Score on the Negative Reactions Scale from the Revised Memory and Behavior Problem Checklist. The scale measures the caregiver's level of reaction to a series of potential problematic behaviors on a 0-4 likert scale; higher numbers indicate a greater degree of distress. The range is 0-96.
Time Frame: baseline to end of treatment (6 months)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Caregiver Website | Caregiver Phone Calls
Number analyzed (Participants) | 20 | 20
units on a scale
  baseline | 16.04 (3.00) | 19.09 (3.08)
  end-of-treatment (6 months) | 20.23 (3.38) | 20.08 (3.57)
Statistical Analysis 1: Comparison: Caregiver Website vs Caregiver Phone Calls; intent to treat analysis; Test type: Superiority or Other; p = .49, Mixed Models Analysis — t test for differential change over time in the two groups t(29)=.70

5. Primary Outcome: Change in Caregiver Depression From Baseline
Description: Total score on the Beck Depression Inventory. The Beck Depression Inventory is a 21 item likert scale instrument with a total range of 0 to 63. Higher scores are indicative of increased endorsement of depressive symptoms. Additionally, it utilizes a cutoff score of13 to indicate probable depression
Time Frame: baseline to end-of-treatment (6 months)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Caregiver Website | Caregiver Phone Calls
Number analyzed (Participants) | 19 | 21
units on a scale
  baseline | 9.27 (1.54) | 9.20 (1.63)
  end of treatment | 8.61 (1.73) | 9.43 (1.83)
Statistical Analysis 1: Comparison: Caregiver Website vs Caregiver Phone Calls; intent to treat analysis; Test type: Superiority or Other; p = .67, Mixed Models Analysis — t test for differential change over time in the two groups t(29)=.43

6. Other Pre Specified Outcome: Number of Participants Placed in Assisted Living or Nursing Homes 12 Months From Baseline
Description: Frequency count of individuals placed in assisted living or nursing homes
Time Frame: baseline to end-of-follow-up (12 months from baseline)
Population: Numbers vary; patients only at risk for out-of-home placement if alive and with data during follow-up periods
Measure: Number; unit: participants
Arm/Group | Caregiver Website | Caregiver Phone Calls
Number analyzed (Participants) | 18 | 16
participants | 2 | 3
Statistical Analysis 1: Comparison: Caregiver Website vs Caregiver Phone Calls; Test type: Superiority or Other; p = .64, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline through 12 months
Arm/Group | Caregiver Website Support | Caregiver Brief Supportive Phone Calls
Serious Adverse Events (participants affected / at risk) | 4/29 | 5/24
Other Adverse Events (participants affected / at risk) | 0/29 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caregiver Website Support (N=29) | Caregiver Brief Supportive Phone Calls (N=24)
fatal (Nervous system disorders) | 3 (3) | 4 (4) — Participants were diagnosed with Alzheimer or other dementia
Hospitalization (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes